CLINICAL TRIAL: NCT05523752
Title: Placement of Four Different Supraglottic Airway Devices by Medicine Faculty Students: A Manikin Study
Brief Title: Insertion of Different Supraglottic Airway Devices on Manikin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Keziban Bollucuoglu, anesthesiologist, Zonguldak Bulent Ecevit University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2022/03-13
Record Dates: First submitted 2022-08-16; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Ventilation; Airway Management; Education
Keywords: Airway management; Supraglottic airway devices; Manikin study; education
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Proseal Laryngeal Mask (Other)
  Interventions: Device: Proseal Laryngeal Mask
- Classic Laryngeal Mask (Other)
  Interventions: Device: Classic Laryngeal Mask
- I-gel (Other)
  Interventions: Device: I-gel
- Suprema Laryngeal Mask (Other)
  Interventions: Device: Suprema Laryngeal Mask

INTERVENTIONS:
Device: Proseal Laryngeal Mask — insertion of Proseal Laryngeal Mask
  Arms: Proseal Laryngeal Mask
Device: Classic Laryngeal Mask — insertion of Classic Laryngeal Mask
  Arms: Classic Laryngeal Mask
Device: I-gel — insertion of I-gel
  Arms: I-gel
Device: Suprema Laryngeal Mask — insertion of Suprema Laryngeal Mask
  Arms: Suprema Laryngeal Mask

SUMMARY:
When tracheal intubation and face mask ventilation fail, and the insertion of supraglottic airway devices (SHA) can provide ventilation, protecting the patient from hypoxemia. Supraglottic airway devices have become an important part of difficult airway algorithms. The European Resuscitation Council Guidelines recommend supraglottic airway devices for airway management by non-specialized healthcare providers. Education through simulators contributes to the development of students without direct contact with patients. In this study, it was aimed to compare the success of placement of four different supraglottic airway devices on the manikin of term 5 students who participate to the Anesthesiology and Reanimation internship.

ELIGIBILITY:
Inclusion Criteria:

* Studying in medical school in term 5
* To have completed anesthesiology and reanimation internship

Exclusion Criteria:

* who do not want to participate in the study
* Students with previous experience with four airway devices

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
difficulty of attempts | during insertion procedure
  pointing the difficulty of insertion from 0 to 100

SECONDARY OUTCOMES:
Time of attempts | during insertion procedure
  time from insertion to ventilation
number of attempts | during insertion procedure
  number of attempts for successfull placement

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes